CLINICAL TRIAL: NCT01135186
Title: Kuvan® (Sapropterin Dihydrochloride) for Improving Gastric Accommodation in Women With Diabetic Gastroparesis (KIGA-DG)
Brief Title: Impact of KUVAN® on Gastric Relaxation in Women With Diabetic Gastroparesis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Linda Nguyen, Principle Investigator, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SU-03252010-5462
Record Dates: First submitted 2010-05-28; First posted 2010-06-02 (Estimated); Results first posted 2017-03-29 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Gastroparesis
MeSH Terms: conditions — Gastroparesis | interventions — sapropterin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sapropterin (Other): open label study of sapropterin dihydrochloride
  Interventions: Drug: sapropterin dihydrochloride

INTERVENTIONS:
Drug: sapropterin dihydrochloride — sapropterin dihydrochloride: 10mg/kg/day
  Other Names: KUVAN

SUMMARY:
Kuvan® (sapropterin dihydrochloride) for Improving Gastric Accommodation in Women with Diabetic Gastroparesis (KIGA-DG)

DETAILED DESCRIPTION:
Patients are invited to participate in a research study of Kuvan® (sapropterin dihydrochloride). We hope to learn whether treatment with Kuvan® is safe and effective in improving the ability of the stomach to relax after eating and improving the symptoms of diabetic gastroparesis. Women are selected as a possible participant in this study because they have diabetes and moderate to severe gastroparesis (meaning stomach empties slowly).

ELIGIBILITY:
Inclusion Criteria:Inclusion Criteria

Patients with moderate to severe symptoms of diabetic gastroparesis will be studied (GCSI >21). Patients should not have post-surgical gastroparesis or dyspeptic symptoms with normal gastric emptying. In order to qualify for inclusion in the trial, patients must satisfy the following inclusion criteria:

1. Diagnosis of diabetes mellitus > 5 years requiring medical therapy
2. Female gender
3. Ages 18-65 years
4. Documentation of delayed gastric emptying on gastric emptying scintigraphy (within 2 years of enrollment)
5. Symptoms of gastroparesis for at least 6 months with Gastroparesis Cardinal Symptom Index (GCSI) score > 21 indicating moderate to severe symptoms
6. Recent negative upper endoscopy or upper GI series within 2 years of enrollment (no evidence of mechanical obstruction or peptic ulcer disease)

Exclusion Criteria:Exclusion Criteria

Patients who satisfy any of the following exclusion criteria will be ineligible for enrollment in the study:

1. Diabetes diagnosed < 5 years prior to the study
2. Male gender
3. Normal gastric emptying
4. Gastroparesis from post-surgical etiologies
5. Another active disorder, which could explain symptoms in the opinion of the investigator
6. Pregnancy
7. History of significant cardiac arrhythmias and/or prolonged QTc
8. Daily use of narcotic analgesics for abdominal pain
9. Contraindications to gastric emptying breath test: patients with a known allergy to egg, wheat, or algae.
10. Underlying seizure disorder
11. Known history of cardiac ischemia
12. Recent clinically significant gastrointestinal bleeding
13. Patients taking Levodopa
14. Any other condition, which in the opinion of the investigator would impede compliance or hinder the completion of the study
15. Failure to give informed consent
16. Surgery for placement of a gastric stimulator within the past 6 months (patients > 6 months post-op with persistent symptoms and delayed gastric emptying are eligible).
17. A normal upper endoscopy not performed within 2 year of study entry.
18. Patients taking phosphodiesterase inhibitors such as sildenafil, vardenafil, tadalafil
19. Patients with renal impairment (i.e. Creatinine > 2.5 mg/dL)
20. Patients with hepatic dysfunction (i.e. ALT and AST values > 2.5x ULN and T. bilirubin > 1.5x ULN)
21. Patients with uncontrolled diabetes, such as HbA1c > 10 mg/dl at screening/baseline will be excluded.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2010-05; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda A Nguyen, Principal Investigator — Stanford University; Pankaj Jay Pasricha, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Background] Soykan I, Sivri B, Sarosiek I, Kiernan B, McCallum RW. Demography, clinical characteristics, psychological and abuse profiles, treatment, and long-term follow-up of patients with gastroparesis. Dig Dis Sci. 1998 Nov;43(11):2398-404. doi: 10.1023/a:1026665728213. PMID 9824125
- [Background] Bell RA, Jones-Vessey K, Summerson JH. Hospitalizations and outcomes for diabetic gastroparesis in North Carolina. South Med J. 2002 Nov;95(11):1297-9. PMID 12539997
- [Background] Stacher G. Diabetes mellitus and the stomach. Diabetologia. 2001 Sep;44(9):1080-93. doi: 10.1007/s001250100619. PMID 11596661
- [Background] Gangula PR, Maner WL, Micci MA, Garfield RE, Pasricha PJ. Diabetes induces sex-dependent changes in neuronal nitric oxide synthase dimerization and function in the rat gastric antrum. Am J Physiol Gastrointest Liver Physiol. 2007 Mar;292(3):G725-33. doi: 10.1152/ajpgi.00406.2006. PMID 17347455
- [Background] Werner ER, Gorren AC, Heller R, Werner-Felmayer G, Mayer B. Tetrahydrobiopterin and nitric oxide: mechanistic and pharmacological aspects. Exp Biol Med (Maywood). 2003 Dec;228(11):1291-302. doi: 10.1177/153537020322801108. PMID 14681545
- [Background] Smirnova VI, Gridchik IE, Tregubenko AD, Khachaturova EA. [Analgesia and intensive therapy during hemicorporectomy]. Anesteziol Reanimatol. 1991 Sep-Oct;(5):46-8. Russian. PMID 1767961

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 9 women with moderate to severe gastroparesis were enrolled at medical clinic.
Groups:
- Open Label Study: sapropterin dihydrochloride
  sapropterin dihydrochloride: sapropterin dihydrochloride: 10mg/kg/day
Period: Overall Study
Arm/Group | Open Label Study
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Open Label Study: sapropterin dihydrochloride
  sapropterin dihydrochloride: sapropterin dihydrochloride: 10mg/kg/day (week 1 through week 4)
  sapropterin dihydrochloride: sapropterin dihydrochloride: 20mg/kg/day (week 5 through week 8)
Arm/Group | Open Label Study
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.56 (15.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Gastric Accommodation
Description: Gastric Accommodation refers to the reflexive relaxation of the upper stomach after swallowing as measured by the Satiety Test at baseline, 4 weeks, and 8 weeks.
  Increased gastric accommodation is considered a positive outcome.
Time Frame: Baseline, 4 Weeks, 8 Weeks
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Open Label Study
Number analyzed (Participants) | 9
ml
  Baseline | 322.22 (137.18)
  4 Weeks | 402.78 (197.03)
  8 Weeks | 450.63 (301.50)

2. Secondary Outcome: Secondary Outcome Measures Will Include Change in Symptom Severity.
Description: Change in symptom severity over the past 2 weeks as measured by the patient reported Gastroparesis Cardinal Symptom Index (GCSI)
  The GCSI is composed of 9 questions.
  Each question asks about symptom severity on a scale of 1-5 listed below.
  0=None 1= Very mild 2= Mild 3=Moderate 4=Severe 5= Very severe
  The 9 scores are summed together for cumulative GCSI score. The minimum cumulative score is '"0" and the maximum cumulative score is "45."
  Once we calculated the cumulative score for each participant, we took the average of all participants cumulative scores giving us the sample mean. This was done at baseline, week 4, and week 8.
  Higher total scores indicate higher symptom severity. Lower total scores indicate lower symptom severity.
Time Frame: Baseline, 4 Weeks, 8 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Open Label Study: sapropterin dihydrochloride
  sapropterin dihydrochloride: sapropterin dihydrochloride: 10mg/kg/day week 1-4, 20mg/kg/day week 5-8.
Arm/Group | Open Label Study
Number analyzed (Participants) | 9
units on a scale
  Baseline | 32.00 (8.67)
  4 Weeks | 23.25 (13.91)
  8 Weeks | 23.67 (13.91)

3. Secondary Outcome: Secondary Outcome Measures Will Include Change in Quality of Life.
Description: Quality of life as impacted by patients with upper gastrointestinal disorders (PAGI-QOL)
  The PAGI-QOl is composed of 30 questions.
  Each question asks about the degree to which a patient's quality of life is impacted by upper gastrointestinal disorders.
  Questions measure quality of life impact on a scale of 1-5 listed below.
  0=none of the time, 1=a little of the time, 2=some of the time, 3=a good bit of the time, 4= most of the time, 5= all of time
  The 30 items are summed together for a cumulative PAGI-QOL score. The minimum cumulative score is "0" and the maximum score is "150."
  Once we calculated the cumulative score for each participant, we took the average of all participants cumulative scores giving us the sample mean. This was done at baseline, week 4, and week 8.
  Lower scores indicate an improved overall quality of life. Higher scores indicate a diminished overall quality of life.
Time Frame: Baseline, 4 Weeks, 8 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Open Label Study: sapropterin dihydrochloride
  sapropterin dihydrochloride: sapropterin dihydrochloride: 10mg/kg/day weeks (1-4) and 20mg/kg/days weeks (week 5-8)
Arm/Group | Open Label Study
Number analyzed (Participants) | 9
units on a scale
  Baseline | 91.22 (28.27)
  4 Weeks | 61.29 (37.83)
  8 Weeks | 60.50 (40.90)

4. Secondary Outcome: Secondary Outcome Measures Will Include Change in Symptom Severity as Measured by the Patient Assessment of Gastrointestinal Disorder-Symptom Severity Index Disorders Symptom Severity Index (PAGI-SYM)
Description: Symptom severity as measured by the Patient Assessment of Upper Gastrointestinal Disorder- Symptom Severity Index. (PAGI-SYM)
  The PAGI-SYM is compose of 20 questions.
  Each question can be answered on a scale of 1-5 (below)
  0 = none, 1=very mild, 2=mild, 3=moderate, 4=severe, 5=very severe
  Cumulative scores were calculated by summing all 20 questions.
  The minimum cumulative scores would be "0" while the maximum cumulative score would be "100"
  Once we calculated the cumulative score for each participant, we took the average of all the cumulative scores giving us the sample mean. This was done at baseline, week 4, and week 8.
  Lower score indicates decreased symptom severity. Higher score indicates increased symptom severity.
Time Frame: Baseline, 4 Weeks, 8 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open Label Study
Number analyzed (Participants) | 9
units on a scale
  Baseline | 54.89 (17.14)
  4 Weeks | 41.50 (23.08)
  8 Weeks | 34.50 (19.71)

ADVERSE EVENTS:
Groups:
- Open Label Study: sapropterin dihydrochloride
  sapropterin dihydrochloride: sapropterin dihydrochloride: 10mg/kg/day (week 1-4) 20 mg/kg/day (week 5-8)
Arm/Group | Open Label Study
Serious Adverse Events (participants affected / at risk) | 1/9
Other Adverse Events (participants affected / at risk) | 0/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label Study (N=9)
Hospitalization for gastroparesis flareup (Gastrointestinal disorders) | 1 (1) — 1 participant was hospitalized for a gastroparesis flare determined not to be related to the study drug. Pt. stopped drug and was given alternative treatment.

LIMITATIONS AND CAVEATS:
A larger sample size is required to confirm the efficacy of saproptetin in increasing gastric accommodation and decreasing gastroparesis symptoms. This would assist in optimal dosing and duration of therapy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No